CLINICAL TRIAL: NCT03852433
Title: A Multicenter, Open-label, Randomized Phase 2b Clinical Study to Assess Efficacy and Safety of Bulevirtide in Combination With Pegylated Interferon Alfa-2a in Patients With Chronic Hepatitis Delta
Brief Title: Study to Assess Efficacy and Safety of Bulevirtide in Combination With Pegylated Interferon Alfa-2a in Participants With Chronic Hepatitis Delta (CHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR204; 2019-001485-15 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Hepatitis Delta
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — bulevirtide; myrcludex-B; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Pegylated Interferon alfa-2a (PEG-IFN alfa) (Active Comparator): Participants will receive PEG-IFN alfa 180 microgram (mcg) once a week subcutaneously for 48 weeks with additional 48 weeks follow-up.
  Interventions: Drug: Peginterferon Alfa-2a (PEG-IFN alfa)
- Bulevirtide 2 mg/day + PEG-IFN alfa (Experimental): Participants will receive bulevirtide 2 mg once a day subcutaneously incombination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 2 mg once a day for 48 weeks and additional 48 weeks follow-up.
  Interventions: Drug: Bulevirtide; Drug: Peginterferon Alfa-2a (PEG-IFN alfa)
- Bulevirtide 10 mg/day + PEG-IFN alfa (Experimental): Participants will receive bulevirtide 10 mg once a day subcutaneously in combination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 10 mg once a day for 48 weeks and additional 48 weeks follow-up.
  Interventions: Drug: Bulevirtide; Drug: Peginterferon Alfa-2a (PEG-IFN alfa)
- Bulevirtide 10 mg once a day (Experimental): Participants will receive bulevirtide 10 mg once a day subcutaneously for 96 weeks with additional 48 weeks follow-up
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — Administered via subcutaneous injections
  Other Names: Myrcludex B; Hepcludex®
  Arms: Bulevirtide 10 mg once a day; Bulevirtide 10 mg/day + PEG-IFN alfa; Bulevirtide 2 mg/day + PEG-IFN alfa
Drug: Peginterferon Alfa-2a (PEG-IFN alfa) — Administered via subcutaneous injections
  Arms: Bulevirtide 10 mg/day + PEG-IFN alfa; Bulevirtide 2 mg/day + PEG-IFN alfa; Pegylated Interferon alfa-2a (PEG-IFN alfa)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of bulevirtide in combination with pegylated interferon in participants with chronic hepatitis delta (CHD).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Positive serum hepatitis delta virus (HDV) antibody results or polymerase chain reaction (PCR) results for serum/ plasma HDV ribonucleic acid (RNA )for at least 6 months before screening.
* Positive PCR results for serum/ plasma HDV RNA at screening.
* Alanine transaminase level >1 x upper limit of normal (ULN), but less than 10 x ULN.
* Serum albumin >28 g/L.
* Thyroid stimulating hormone (TSH) within normal ranges (including on medication for control of thyroid function)
* Negative urine pregnancy test for females of childbearing potential.
* Inclusion criteria for female individuals:

  * Postmenopausal for at least 2 years, or
  * Surgically sterile (total hysterectomy or bilateral oophorectomy, bilateral tubal ligation, staples, or another type of sterilization), or
  * Abstinence from heterosexual intercourse throughout the treatment period, or
  * Willingness to use highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive) throughout the treatment period and for 6 months after the last dose of the study medication.
* Male individuals must agree to use a highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive used by female partners) and not to donate sperm throughout the treatment period and for 6 months after the last dose of the study medication.

Exclusion Criteria:

* Child-Pugh hepatic insufficiency score of B-C or over 6 points. Note: Child-Pugh hepatic insufficiency score of 6 points is allowed. Only individuals with compensated cirrhosis are allowed. Uncomplicated oesophageal varices allowed; individuals with current bleeding or ligation, or history of bleeding or ligation within the last 2 years are excluded.
* Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) coinfection. Individuals with HCV antibodies can be enrolled, if screening HCV RNA test is negative.
* Creatinine clearance < 60 mL/min as estimated using Cockcroft-Gault formula.
* Total bilirubin ≥ 34.2 µmol/L. (Individuals with higher total bilirubin values may be included after the consultation with the Study Medical Monitor, if such elevation can be clearly attributed to Gilbert's syndrome associated with low-grade hyperbilirubinemia.)
* Evidence of an active or suspected malignancy, or an untreated pre-malignancy disorder, or a history of malignancy within the last 5 years (with the exception of successfully treated carcinoma of the cervix in situ and successfully treated basal cell carcinoma and squamous cell carcinoma not less than 1 year prior to screening [and no more than 3 excised skin cancer within the last 5 years prior to screening]) or history of hepatic carcinoma.
* Systemic connective tissue disorders.
* New York Heart Association (NYHA) class III-IV congestive heart failure.
* Individuals with uncontrolled arterial hypertension: systolic blood pressure > 150 mm Hg and/ or diastolic blood pressure > 100 mm Hg at Screening.
* Previous or unstable concurrent diseases or conditions that prevent individual's enrolment into the study.
* Individuals with mental disorders or social circumstances that preclude them from following protocol requirements.
* Current or previous decompensated liver disease, including coagulopathy, hepatic encephalopathy and esophageal varices hemorrhage.
* One or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.). Gilbert's syndrome, a benign disorder associated with low-grade hyperbilirubinemia, will not exclude individauls from participation in this trial. Autoimmune hepatitis stigmata attributed to HDV infection in the opinion of the investigator are allowed.
* White blood cells (WBC) count < 3000 cells/mm^3 (<1500 if African individuals).
* Absolute neutrophil count < 1500 cells/mm^3 (<1000 if African individuals).
* Platelet count < 90,000 cells/mm^3.
* Haemoglobin < 12 g/dL.
* Use of prohibited psychotropic agents at Screening.
* Use of interferons within 6 months before Screening.
* History of solid organ transplantation.
* Current alcohol abuse or alcohol abuse within 6 months prior to enrolment in this study; current drug addict or history of drug use within 2 years prior to Screening.
* History of disease requiring regular use of systemic glucocorticosteroids (inhalative glucocorticosteroids are allowed) or other immunosuppressants.
* Pregnant or breast-feeding females.
* Participation in another clinical study with investigational drugs within 30 days prior to randomization.
* Receipt of bulevirtide previously, e.g. in clinical trials.
* Inability to follow protocol requirements and undergo all protocol procedures. Note: Individuals with medical contraindication for liver biopsy are allowed to participate in this study. Such individuals will exempt from liver biopsy requirements in this study. Individuals receiving prohibited treatment at screening cannot be included into the study unless this treatment is withdrawn prior to randomization.
* Contraindications, intolerance or hypersensitivity to interferons alfa, genetically engineered E.coli medications, polyethylene glycol or other components of peginterferon alfa-2а.
* Presence or history of severe retinopathy, significant diabetic or hypertensive retinopathy.
* Uncontrolled diabetes mellitus.
* Uncontrolled cardiovascular disorders within 6 months before screening.
* History of autoimmune disorder (e.g. myositis, hepatitis, thrombotic thrombocytopenic purpura, idiopathic thrombocytopenic purpura, severe psoriasis, rheumatoid arthritis, interstitial nephritis, thyroiditis, and systemic lupus erythematosus)
* Presence or history of significant psychiatric disorder (e.g. severe depression, suicide attempt, severe neurosis or cognitive disorder).
* Presence or history of chronic lung disease with respiratory malfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Medical Monitor, Study Chair — Gilead Sciences
Locations (20):
- France (6):
  - Hôpital Beaujon-Pavillon Abrami -Sce Hépatologie, Clichy
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Hospital Croix Rousee, Lyon
  - Hôpital Saint Joseph Hépato-Gastroentérologie, Marseille
  - CH Pitié-Salpétrière - Hépato-Gastroentérologie, Paris
  - Hôpital Cochin - Unité d'Hépatologie Pavillon Achard, Paris
- Moldova (2):
  - Infectious Clinical Hospital "T. Ciorba", Department 4 / Medical University Department of Infectious Diseases, Chisinau
  - Infectious Clinical Hospital "T. Ciorba", Department 5 / Medical University Department of Infectious Diseases, Chisinau
- Romania (4):
  - "Matei Bals" National Institute of Infectious Diseases, Hospital department, Bucharest
  - "Matei Bals" National Institute of Infectious Diseases,Clinical Trials department, Bucharest
  - "Victor Babes" Centre of Diagnostic and Treatment, Bucharest
  - Dr. V. Babes Clinical Hospital of Infectious and Tropical Diseases, Bucharest
- Russia (8):
  - State Budgetary Educational Institution of Higher Professional Education "South Ural State Medical University" of the Ministry of Healthcare of the Russian Federation, Chelyabinsk
  - Specialized clinical Infectious diseases Hospital, Krasnodar
  - Federal Budget Institute of Science "Central Research Institute for Epidemiology" of Federal Service on Consumers Rights Protection and Human Well-Being Surveillance, Moscow
  - Federal State Budgetary Institution National Research Medical Center for Phthisiopulmonology and Infectious Diseases of the Ministry of Health of the Russian Federation, Moscow
  - LLC"Clinic of Modern Medicine", Moscow
  - Moscow Regional Scientific and Research Clinical Institute, Moscow
  - N.V.Sklifosovsky Scientific Research Institute of Emergency care of the Moscow Healthcare Department, Moscow
  - LLC Medical Company "Hepatolog", Samara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asselah T, Arama SS, Bogomolov P, Bourliere M, Fontaine H, Gherlan GS, et al. Safety and Efficacy of Bulevirtide Monotherapy and in Combination with Peginterferon Alfa-2a in Patients with Chronic Hepatitis Delta: 24 Weeks Interim Data of MYR204 Phase 2b Study [Presentation]. European Association for the Study of the Liver (EASL): The Digital International Liver Congress; 2021 23-26 June.
- [Background] Asif B, Koh C. Hepatitis D virus (HDV): investigational therapeutic agents in clinical trials. Expert Opin Investig Drugs. 2022 Sep;31(9):905-920. doi: 10.1080/13543784.2021.1977795. Epub 2021 Oct 1. PMID 34482769
- [Background] Soriano V, Moreno-Torres V, Trevino A, Corral O, de Mendoza C. Bulevirtide in the Treatment of Hepatitis Delta: Drug Discovery, Clinical Development and Place in Therapy. Drug Des Devel Ther. 2023 Jan 21;17:155-166. doi: 10.2147/DDDT.S379964. eCollection 2023. PMID 36712949
- [Background] Asselah T, Lampertico P, Wedemeyer H, Streinu-Cercel A, Pantea V, Lazar S, et al. Efficacy and Safety of Bulevirtide in Combination with Pegylated Interferon alfa-2a in Patients with Chronic Hepatitis Delta: Primary Endpoint Results from a Phase 2b Open-Label, Randomized, Multicenter Study MYR204. [Poster #5009]. AASLD - The Liver Meeting; 2023 November 10-24; Boston, MA.
- [Derived] Asselah T, Lampertico P, Aleman S, Bourliere M, Streinu-Cercel A, Bogomolov P, Morozov V, Stepanova T, Lazar S, Manuilov D, Mercier RC, Tseng S, Ye L, Flaherty JF, Osinusi A, Da BL, Chee GM, Lau AH, Brunetto MR, Wedemeyer H. Bulevirtide Monotherapy Is Safe and Well Tolerated in Chronic Hepatitis Delta: An Integrated Safety Analysis of Bulevirtide Clinical Trials at Week 48. Liver Int. 2025 Apr;45(4):e16174. doi: 10.1111/liv.16174. Epub 2024 Dec 8. PMID 39648559
- [Derived] Asselah T, Chulanov V, Lampertico P, Wedemeyer H, Streinu-Cercel A, Pantea V, Lazar S, Placinta G, Gherlan GS, Bogomolov P, Stepanova T, Morozov V, Syutkin V, Sagalova O, Manuilov D, Mercier RC, Ye L, Da BL, Chee G, Lau AH, Osinusi A, Bourliere M, Ratziu V, Pol S, Hilleret MN, Zoulim F. Bulevirtide Combined with Pegylated Interferon for Chronic Hepatitis D. N Engl J Med. 2024 Jul 11;391(2):133-143. doi: 10.1056/NEJMoa2314134. Epub 2024 Jun 6. PMID 38842520
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=MYR%20204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the France, Moldova, Romania and Russia.
Pre-assignment Details: 258 participants were screened. Participants were assigned to arms A: Pegylated Interferon Alfa-2a (PEG-IFN Alfa), B: Bulevirtide 2 mg/Day + PEG-IFN Alfa, C: Bulevirtide 10 mg/Day + PEG-IFN Alfa and D: Bulevirtide 10 mg/Day to the respective treatment.
Groups:
- Pegylated Interferon Alfa-2a (PEG-IFN Alfa): Participants received PEG-IFN alfa 180 microgram (mcg) once a week subcutaneously for 48 weeks with additional 48 weeks follow-up.
- Bulevirtide 2 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 2 mg once a day subcutaneously in combination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 2 mg once a day for 48 weeks and additional 48 weeks follow-up.
- Bulevirtide 10 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 10 mg once day subcutaneously in combination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 10 mg once a day for 48 weeks and additional 48 weeks follow-up.
  .
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg once day subcutaneously for 96 weeks with additional 48 weeks follow-up.
Period: Overall Study
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Started | 25 | 50 | 50 | 50
Completed | 17 | 38 | 45 | 45
Not Completed | 8 | 12 | 5 | 5
Not completed — Withdrawal of consent | 5 | 8 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Randomized but never treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Analysis Set included all participants who were enrolled (informed consent signed) and randomized in the study.
Groups:
- Bulevirtide 10 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 10 mg once a day subcutaneously in combination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 10 mg once a day for 48 weeks and additional 48 weeks follow-up.
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg once a day subcutaneously for 96 weeks with additional 48 weeks follow-up.
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day | Total~(N=174)
Number analyzed (Participants) | 25 | 50 | 50 | 50 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 50 | 49 | 50 | 174
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (8.2) | 41 (9.3) | 41 (8.6) | 40 (8.5) | 41 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 15 | 12 | 50
  Male | 19 | 33 | 35 | 38 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 4 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 2 | 7
  White | 21 | 44 | 43 | 44 | 152
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity data was not collected in this study.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 14 | 29 | 22 | 27 | 92
  Romania | 6 | 11 | 12 | 12 | 41
  Moldova | 3 | 7 | 12 | 9 | 31
  France | 2 | 3 | 4 | 2 | 11
HDV RNA [Mean (Standard Deviation); unit: log10 IU/mL] — Full Analysis Set included all randomized participants who took at least 1 dose of study drug.
  log10 IU/mL | 5.20 (1.064) | 5.27 (1.355) | 5.09 (1.343) | 5.45 (1.098) | 5.26 (1.242)
Liver Stiffness [Mean (Standard Deviation); unit: kPa] — Participants from Full Analysis Set with available data were analyzed.
  kPa | 15.8 (11.57) | 12.8 (6.43) | 12.5 (7.60) | 12.7 (6.65) | 13.1 (7.72)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response at Week 24 After the Scheduled End of Treatment (SVR24)
Description: SVR24 was defined as undetectable hepatitis delta virus (HDV) RNA (HDV RNA value < lower limit of quantitation [LLOQ] with target not detected) at 24 weeks after the scheduled end of treatment (EOT).
Time Frame: 24 weeks after EOT (Week 72 for Arm A and study Week 120 for Arms B, C, and D)
Population: Full Analysis Set, is defined as all randomized participants who received at least 1 dose of study drug (Peg-IFNα and/or BLV).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 24 | 50 | 50 | 50
percentage of participants | 16.7 [4.7 to 37.4] | 32.0 [19.5 to 46.7] | 46.0 [31.8 to 60.7] | 12.0 [4.5 to 24.3]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0003, Fisher Exact; Difference in percentages = 34.0, 95% CI 2-sided [14.6 to 50.4]
Statistical Analysis 2: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 2 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.2631, Fisher Exact; Difference in percentages = 15.3, 95% CI 2-sided [-8.2 to 34.2]
Statistical Analysis 3: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.0197, Fisher Exact; Difference in percentages = 29.3, 95% CI 2-sided [1.8 to 48.2]
Statistical Analysis 4: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.7186, Fisher Exact; Difference in percentages = -4.7, 95% CI 2-sided [-26.3 to 11.8]
Statistical Analysis 5: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.2184, Fisher Exact; Difference in percentages = 14.0, 95% CI 2-sided [-5.5 to 32.7]
Statistical Analysis 6: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0283, Fisher Exact; Difference in percentages = -20.0, 95% CI 2-sided [-36.1 to -3.5]

2. Secondary Outcome: Percentage of Participants With Undetectable HDV RNA at Week 48
Description: Undetectable HDV RNA at Week 48 means undetectable (< LLOQ, target not detected) HDV RNA at Week 48.
Time Frame: Week 48
Population: Participants from Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 24 | 50 | 50 | 50
percentage of participants | 20.8 [7.1 to 42.2] | 40.0 [26.4 to 54.8] | 60.0 [45.2 to 73.6] | 10.0 [3.3 to 21.8]

3. Secondary Outcome: Percentage of Participants With Undetectable HDV RNA at Week 96 (Arms B, C, and D Only)
Description: Undetectable HDV RNA at Week 96 means undetectable (< LLOQ, target not detected) HDV RNA at Week 96.
Time Frame: Week 96
Population: Participants from Full Analysis Set were analyzed. Per prespecified analysis, the data for this outcome measure was collected only for Arms B, C, and D at the scheduled Week 96 visit. Hence the data for Arm A is not reported for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants | 44.0 [30.0 to 58.7] | 70.0 [55.4 to 82.1] | 22.0 [11.5 to 36.0]

4. Secondary Outcome: Percentage of Participants With Combined Response at Week 24 After the Scheduled End of Treatment
Description: Combined response was defined as fulfilment of 2 conditions simultaneously: 1) undetectable HDV RNA or decrease by ≥ 2 log10 IU/mL from baseline, alanine aminotransferase (ALT) normalization, defined as an ALT value within the normal range, based on the central laboratories [Russian sites: ≤ 31 U/L for females and ≤ 41 U/L for males; all other sites: ≤ 34 U/L for females and ≤ 49 U/L for males]).
Time Frame: 24 weeks after EOT (Week 72 for Arm A and Week 120 for Arms B, C, and D)
Population: Participants from Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bulevirtide 10 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 10 mg once a day subcutaneously in combination with PEG-IFN alfa 180 mcg once a week subcutaneously for 48 weeks followed by bulevirtide 10 mg once a day for 48 weeks and additional48 weeks follow-up
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 24 | 50 | 50 | 50
percentage of participants | 20.8 [7.1 to 42.2] | 36.0 [22.9 to 50.8] | 52.0 [37.4 to 66.3] | 26.0 [14.6 to 40.3]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0134, Fisher Exact; Difference in percentages = 26.0, 95% CI 2-sided [6.0 to 44.0]

5. Secondary Outcome: Percentage of Participants With Combined Response at Week 48 After the Scheduled End of Treatment
Description: Combined response is defined as fulfilment of 2 conditions simultaneously: 1) undetectable HDV RNA or decrease by ≥ 2 log10 IU/mL from baseline, ALT normalization, defined as an ALT value within the normal range, based on the central laboratories [Russian sites: ≤ 31 U/L for females and ≤ 41 U/L for males; all other sites: ≤ 34 U/L for females and ≤ 49 U/L for males]).
Time Frame: 48 weeks after EOT (Week 96 for Arm A and Week 144 for Arm B, C, and D)
Population: Participants from Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 24 | 50 | 50 | 50
percentage of participants | 33.3 [15.6 to 55.3] | 32.0 [19.5 to 46.7] | 46.0 [31.8 to 60.7] | 18.0 [8.6 to 31.4]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0049, Fisher Exact; Difference in percentages = 28.0, 95% CI 2-sided [8.2 to 45.1]

6. Secondary Outcome: Percentage of Participants With Sustained Virological Response 48 After the Scheduled End of Treatment (SVR 48)
Description: SVR 48 is defined as undetectable hepatitis delta virus (HDV) RNA (HDV RNA value < lower limit of quantitation [LLOQ] with target not detected) at 48 weeks after the scheduled end of treatment.
Time Frame: 48 weeks after EOT (Week 96 for Arm A; Week 144 for Arms B, C, and D)
Population: Participants from Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 24 | 50 | 50 | 50
percentage of participants | 25.0 [9.8 to 46.7] | 26.0 [14.6 to 40.3] | 46.0 [31.8 to 60.7] | 12.0 [4.5 to 24.3]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0003, Fisher Exact; Difference in percentages = 34.0, 95% CI 2-sided [14.6 to 50.4]
Statistical Analysis 2: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 2 mg/Day + PEG-IFN Alfa; Test type: Other; p = 1.0000, Fisher Exact; Difference in percentages = 1.0, 95% CI 2-sided [-22.8 to 21.4]
Statistical Analysis 3: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.1265, Fisher Exact; Difference in percentages = 21.0, 95% CI 2-sided [-5.3 to 42.2]
Statistical Analysis 4: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.1863, Fisher Exact; Difference in percentages = -13.0, 95% CI 2-sided [-35.3 to 5.4]
Statistical Analysis 5: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.0601, Fisher Exact; Difference in percentages = 20.0, 95% CI 2-sided [1.0 to 38.2]
Statistical Analysis 6: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.1247, Fisher Exact; Difference in percentages = -14.0, 95% CI 2-sided [-29.9 to 1.7]

7. Secondary Outcome: Change From Baseline in Liver Stiffness as Measured by Elastography at Week 48
Description: The mixed-effects models for repeated measurements (MMRM) model was used for analysis.
Time Frame: Baseline, Week 48
Population: Participants from Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 18 | 45 | 47 | 48
kPa | -0.02 [-2.29 to 2.25] | -1.85 [-3.42 to -0.28] | -1.79 [-3.21 to -0.36] | -3.34 [-4.84 to -1.85]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0717, MMRM; Difference in LS Mean = 1.56, 95% CI 2-sided [-0.14 to 3.26]
Statistical Analysis 2: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 2 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.1563, MMRM; Difference in LS Mean = -1.84, 95% CI 2-sided [-4.39 to 0.71]
Statistical Analysis 3: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.1626, MMRM; Difference in LS Mean = -1.80, 95% CI 2-sided [-4.33 to 0.73]
Statistical Analysis 4: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0099, MMRM; Difference in LS Mean = -3.34, 95% CI 2-sided [-5.87 to -0.82]
Statistical Analysis 5: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.9384, MMRM; Difference in LS Mean = 0.07, 95% CI 2-sided [-1.67 to 1.81]
Statistical Analysis 6: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0875, MMRM; Difference in LS Mean = -1.49, 95% CI 2-sided [-3.20 to 0.22]

8. Secondary Outcome: Change From Baseline in Liver Stiffness as Measured by Elastography at Week 96
Description: The MMRM model was used for analysis.
Time Frame: Baseline, Week 96
Population: Participants from Full Analysis Set with available data were analyzed. Per prespecified analysis, the data for this outcome measure was collected only for Arms B, C, and D at the scheduled Week 96 visit. Hence the data for Arm A is not reported for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 43 | 47 | 46
kPa | -3.37 [-4.94 to -1.80] | -3.70 [-5.11 to -2.29] | -3.85 [-5.35 to -2.35]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.8645, MMRM; Difference in LS Mean = 0.15, 95% CI 2-sided [-1.54 to 1.83]
Statistical Analysis 2: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.7033, MMRM; Difference in LS Mean = -0.33, 95% CI 2-sided [-2.06 to 1.39]
Statistical Analysis 3: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.5806, MMRM; Difference in LS Mean = -0.48, 95% CI 2-sided [-2.18 to 1.23]

9. Secondary Outcome: Change From Baseline in Liver Stiffness as Measured by Elastography at Week 144
Description: The MMRM model was used for analysis.
Time Frame: Baseline, 48 weeks after EOT (Week 96 for Arm A and study Week 144 for Arms B, C, and D)
Population: Participants from Full Analysis Set were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Groups:
- Bulevirtide 10 mg Once a Day: Participants received bulevirtide 10 mg once a day subcutaneously for 96 weeks with additional 48 weeks follow-up.
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg Once a Day
Number analyzed (Participants) | 16 | 32 | 40 | 40
kPa | -0.31 [-2.75 to 2.12] | -2.35 [-4.20 to -0.50] | -2.47 [-4.12 to -0.83] | -0.79 [-2.53 to 0.94]
Statistical Analysis 1: Comparison: Bulevirtide 10 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg Once a Day; Test type: Other; p = 0.1103, MMRM; Difference in LS Mean = -1.68, 95% CI 2-sided [-3.75 to 0.39]
Statistical Analysis 2: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 2 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.1533, MMRM; Difference in LS Mean = -2.05, 95% CI 2-sided [-4.88 to 0.77]
Statistical Analysis 3: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.1129, MMRM; Difference in LS Mean = -2.22, 95% CI 2-sided [-4.98 to 0.53]
Statistical Analysis 4: Comparison: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) vs Bulevirtide 10 mg Once a Day; Test type: Other; p = 0.6753, MMRM; Difference in LS Mean = -0.58, 95% CI 2-sided [-3.34 to 2.17]
Statistical Analysis 5: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg/Day + PEG-IFN Alfa; Test type: Other; p = 0.9124, MMRM; Difference in LS Mean = -0.12, 95% CI 2-sided [-2.28 to 2.04]
Statistical Analysis 6: Comparison: Bulevirtide 2 mg/Day + PEG-IFN Alfa vs Bulevirtide 10 mg Once a Day; Test type: Other; p = 0.1526, MMRM; Difference in LS Mean = 1.56, 95% CI 2-sided [-0.59 to 3.70]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to approximately 144 weeks; Adverse events: Pegylated Interferon Alfa-2a (PEG-IFN Alfa) arm: Week 48 plus 30 days; all other arms: Week 96 plus 30 days
Description: All-cause moratlity: Participants from All Randomized Set with available data were analyzed.
  Adverse events: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Pegylated Interferon Alfa-2a (PEG-IFN Alfa): Participants received PEG-IFN alfa 180 microgram (mcg) once a week for 48 weeks.
- Bulevirtide 2 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 2 mg once a day in combination with PEG-IFN alfa 180 mcg once a week for 48 weeks followed by bulevirtide 2 mg once a day for 48 weeks.
- Bulevirtide 10 mg/Day + PEG-IFN Alfa: Participants received bulevirtide 10 mg once a day in combination with PEG-IFN alfa 180 mcg once a week for 48 weeks followed by bulevirtide 10 mg once a day for 48 weeks.
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg once a day for 96 weeks.
Arm/Group | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) | Bulevirtide 2 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day + PEG-IFN Alfa | Bulevirtide 10 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/50 | 1/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/24 | 3/50 | 8/50 | 2/50
Other Adverse Events (participants affected / at risk) | 22/24 | 49/50 | 50/50 | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) (N=24) | Bulevirtide 2 mg/Day + PEG-IFN Alfa (N=50) | Bulevirtide 10 mg/Day + PEG-IFN Alfa (N=50) | Bulevirtide 10 mg/Day (N=50)
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 1
Covid-19 pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Hepatitis B reactivation (Infections and infestations) | 0 | 0 | 1 | 0
Injection site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa-2a (PEG-IFN Alfa) (N=24) | Bulevirtide 2 mg/Day + PEG-IFN Alfa (N=50) | Bulevirtide 10 mg/Day + PEG-IFN Alfa (N=50) | Bulevirtide 10 mg/Day (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 13 | 26 | 27 | 8
Lymphopenia (Blood and lymphatic system disorders) | 7 | 12 | 15 | 5
Neutropenia (Blood and lymphatic system disorders) | 12 | 23 | 28 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 23 | 24 | 8
Angina pectoris (Cardiac disorders) | 2 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 3 | 2 | 4
Presbyopia (Eye disorders) | 2 | 1 | 0 | 0
Retinal vascular disorder (Eye disorders) | 1 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 4 | 3
Asthenia (General disorders) | 3 | 7 | 6 | 4
Chills (General disorders) | 0 | 4 | 0 | 2
Influenza like illness (General disorders) | 10 | 22 | 20 | 2
Injection site erythema (General disorders) | 0 | 4 | 4 | 4
Injection site reaction (General disorders) | 0 | 5 | 4 | 0
Pyrexia (General disorders) | 5 | 8 | 13 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 1 | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0 | 2 | 4
Covid-19 (Infections and infestations) | 0 | 3 | 5 | 2
Urinary tract infection (Infections and infestations) | 0 | 3 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 6 | 5 | 1
Alanine aminotransferase increased (Investigations) | 8 | 5 | 12 | 5
Alpha-2 macroglobulin increased (Investigations) | 0 | 1 | 3 | 2
Amylase increased (Investigations) | 0 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 8 | 6 | 10 | 3
Bile acids increased (Investigations) | 1 | 1 | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 6 | 2 | 7 | 3
Lipase increased (Investigations) | 1 | 4 | 2 | 4
Neutrophil count decreased (Investigations) | 3 | 11 | 12 | 1
Platelet count decreased (Investigations) | 2 | 9 | 7 | 1
Prothrombin level decreased (Investigations) | 0 | 1 | 3 | 1
Weight decreased (Investigations) | 3 | 3 | 4 | 2
White blood cell count decreased (Investigations) | 2 | 10 | 8 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 9 | 13 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 3 | 2 | 5
Headache (Nervous system disorders) | 2 | 7 | 7 | 7
Anxiety (Psychiatric disorders) | 0 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 4 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03852433/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03852433/SAP_001.pdf